CLINICAL TRIAL: NCT06742541
Title: Spherical Implantable Collamer Lens With Postoperative Adjunctive LASIK in the Treatment of High Compound Hyperopic Astigmatism
Brief Title: ICL and LASIK for Hyperopic Astigmatism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Daniel Li, Resident Physician, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGC81
Record Dates: First submitted 2024-12-10; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Astigmatism; Hyperopia
Keywords: ICL; LASIK; Hyperopia; Astigmatism
MeSH Terms: conditions — Astigmatism; Hyperopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with high compound hyperopic astigmatism (Experimental): eyes with ≥3.50 D hyperopia and ≥2.00 D of astigmatism undergoing planned surgery receiving a spherical Implantable Collamer Lens (ICL) followed by a planned adjunctive LASIK postoperatively
  Interventions: Device: Implantable Collamer Lens (ICL) followed by a planned adjunctive LASIK postoperatively

INTERVENTIONS:
Device: Implantable Collamer Lens (ICL) followed by a planned adjunctive LASIK postoperatively — Planned surgery to receive a spherical Implantable Collamer Lens (ICL) followed by a planned adjunctive LASIK postoperatively
  Other Names: ICL + LASIK

SUMMARY:
This study investigates a two-step treatment for people with severe farsightedness combined with astigmatism. The first step involves implanting a specially designed lens inside the eye (a spherical Implantable Collamer Lens, or ICL) to improve vision. Later, a laser procedure (LASIK) is performed to fine-tune the results for even better clarity.

DETAILED DESCRIPTION:
To assess refractive and visual outcomes of a spherical Implantable Collamer Lens (ICL) followed by planned postoperative adjunctive laser-assisted in situ keratomileusis (LASIK) in the treatment of high compound hyperopic astigmatism. In this prospective, multi-center, multi-surgeon, single-arm study, eyes with ≥3.50 D hyperopia and ≥2.00 D of astigmatism underwent surgery receiving a spherical Implantable Collamer Lens (ICL) followed by a planned adjunctive LASIK postoperatively. Outcomes measures included postoperative uncorrected (UDVA) and corrected distance visual acuity (CDVA), manifest refraction, spherical (SEQ) and defocus equivalent (DEQ), efficacy index, safety index, and astigmatism vector analyses.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative hyperopic sphere of ≥+3.50 D
* Astigmatism of ≥+2.00 D
* Stable refraction for the previous 12 months
* Age older or equal to 18 years
* Anterior chamber depth (ACD) from corneal endothelium to anterior lens capsule of 3.0 mm or greater

Exclusion Criteria:

* Age younger than 18 years
* Patients lost to follow-up
* Cataract formation
* History of glaucoma or retinal detachment
* Macular degeneration
* Diabetic retinopathy
* History of ocular inflammation
* Signifcant irregular corneal topography
* Evidence of inconsistent imaging from dry eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Post-operative visual acuitiy | 90 days after lasik surgery
  postoperative uncorrected (UDVA) and corrected distance visual acuity (CDVA)

SECONDARY OUTCOMES:
Manifest refraction | 90 days after lasik surgery
  The refraction (glasses prescription required) done manually of the operated eye
Spherical (SEQ) and defocus equivalent (DEQ) | 90 days after LASIK surgery
  SEQ: a single value used to describe a refractive error, combining the spherical and cylindrical components of a prescription DEQ: quantifies the overall refractive blur from spherical and cylindrical components
Efficacy Index and Safety Index | 90 days after LASIK surgery
  Efficacy Index: ratio of postoperative uncorrected distance visual acuity (UDVA) to preoperative corrected distance visual acuity (CDVA) Safety Index: ratio of postoperative corrected distance visual acuity (CDVA) to the preoperative CDVA
Astigmatism Vector Analysis | 90 days after LASIK surgery
  The residual astigmatism left after surgery, representing the deviation from the intended correction.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Wallerstein, MD, Principal Investigator — McGill University
Locations (1):
- Vision Group Canada, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No
Small study of only 32 patients, individual data will not be shared to protect patient confidentiality.

REFERENCES:
- [Derived] Li DQ, Gauvin M, Rocha G, Trottier P, Racine L, Wallerstein A. Spherical implantable collamer lens with postoperative adjunctive LASIK in the treatment of high compound hyperopic astigmatism. BMC Ophthalmol. 2025 Jan 24;25(1):44. doi: 10.1186/s12886-024-03828-5. PMID 39856569